CLINICAL TRIAL: NCT00193817
Title: Three Field Radical Esophagectomy Versus Two Field Esophagectomy - a Prospective Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tata Memorial Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMH 111/IM-2004; DAECTC/Projno 5 / 2004-05
Record Dates: First submitted 2005-09-14; First posted 2005-09-19 (Estimated); Last update posted 2006-02-07 (Estimated); Status verified 2005-07

CONDITIONS: Cancer of Esophagus
Keywords: Cancer; Esophagus; Lymphadenectomy
MeSH Terms: conditions — Esophageal Neoplasms; Neoplasms

INTERVENTIONS:
Procedure: Two field vs Three field lymphadenectomy

SUMMARY:
Surgery is the standard treatment for esophageal (food pipe) cancer. Esophageal cancer is known to spread to the lymph nodes (glands) adjacent to the esophagus. The extent of lymph nodes that need to be removed along with removal of the esophagus is a controversial topic. The basic surgery will remain the same i.e., the foodpipe in the chest will be removed and a new substitute will be created from the stomach and joined to the foodpipe in the neck. This will involve incisions in the chest, abdomen and neck. We intend to compare two types of lymphadenectomy (removal of lymph nodes) - the two field lymphadenectomy, whereby the lymph nodes in the abdomen and the lower half of the chest will be removed and three field lymphadenectomy, wherein lymph nodes in the abdomen, the whole chest and the lower neck will be removed. Both these procedures are practised widely worldwide and there is no definite scientific evidence showing the superiority of either of them. We are conducting this study to see whether one of these procedures is superior to the other. Seven hundred patients are expected to participate in this study.

DETAILED DESCRIPTION:
Three field radical esophagectomy versus two field esophagectomy - a prospective randomized controlled trial

Background Esophageal cancer is a common problem worldwide and is associated with poor prognosis. Surgery is the mainstay of treatment and offers the only realistic possibility of cure and long term survival. Neoadjuvant and adjuvant chemotherapy and radiotherapy have been tried in addition to surgery and have only marginally impacted on survival. In spite of advancements in postoperative care and refinements in surgical technique, overall results with surgery have been disappointing. Moreover studies of neoadjuvant and adjuvant therapy have been confounded by the lack of a uniform surgical approach and extent of lymphadenectomy.

The efficacy of prophylactic radical lymph node dissection in surgical treatment of esophageal cancer has been a topic of major controversy for many years. It has not been studied in a randomized controlled trial with adequate numbers. Non randomized studies have been criticized on the basis of selection bias and stage migration. There is presently no convincing evidence regarding improvement in survival by extensive three field lymphadenectomy.

Objectives

1. To compare overall survival after three field and two field esophagectomy
2. To compare locoregional recurrence, disease free survival after three field and two field esophagectomy
3. To compare postoperative morbidity and mortality in the two groups
4. To evaluate short and long term quality of life after the two procedures

Design Prospective randomized controlled trial Setting Tertiary level comprehensive cancer care centre in Western India. Patients and methods All patients with biopsy proven carcinoma of the esophagus presenting to our hospital will be considered for the study.

Inclusion criteria

1. Patients with biopsy or cytology proven (squamous or adenocarcinoma) esophageal cancer (including Siewert's type I and II CO junction cancers)
2. Patients with staging investigations indicating operability
3. Surgical plan for total transthoracic esophagectomy

Exclusion criteria

1. Patients with low performance status (ECOG score > 1)
2. Past history of malignancy
3. Staging investigations indicating advanced disease
4. Patients medically unfit for surgical resection
5. Patients with pulmonary reserve inadequate to undergo thoracotomy and extensive mediastinal dissection
6. Patients considered for salvage surgery after definitive chemoradiotherapy
7. Patients unreliable for follow up
8. Patients above the age of 70 years
9. Patients with enlarged supracarinal nodes on CT scan / EUS
10. Grossly enlarged supracarinal lymph nodes seen intraoperatively
11. Patients with Siewert's type III cancers.

A detailed history including the main complaints and symptoms, symptoms suggestive of advanced disease or dissemination, comorbid conditions and performance status of the patient will be recorded on presentation. A confirmed diagnosis of esophageal carcinoma will be documented in our hospital.

Staging investigations will be standard and will include

1. Computed Tomography (CT) scans in all patients
2. Endoscopic Ultrasonography (EUS) wherever possible
3. Fiberoptic bronchoscopy (all upper and middle third growths and patients with history of recent voice change).
4. Symptomatic patients will undergo further investigations depending on the symptom.

Patients undergoing neoadjuvant chemotherapy or chemoradiotherapy will not be excluded but will be one of the stratification criteria for randomization. Patients will be assessed for operability by a team including two qualified thoracic surgeons and a radiologist. All patients will undergo routine and special investigations where indicated to assess fitness for major surgery and anesthesia. The perioperative risk will be assessed by a combination of the American Society of Anesthesiologists (ASA) grading and a modified risk score (Annexure 1). Patients with ASA grade I or II and those who have low or intermediate risk according to the modified risk scoring system will be considered for the trial. Patients will be explained about the trial and written informed consent will be taken (Annexure 2). Patients considered operable (either per primum or after neoadjuvant therapy) and fit for either procedure and who consent for the trial (Eligibility confirmation and randomization form, annexure 3) will be randomized into two groups.

Randomization Block randomization will be done using a computer generated sheet. Randomization will be performed intraoperatively after confirming resectability of the primary tumor and confirming the absence of grossly enlarged supracarinal lymph nodes

Stratification criteria

1. Preoperative T stage (T1&2, T3 and T4)
2. Preoperative N stage (N0, N1)
3. Level of disease (upper, middle and lower third)
4. Neoadjuvant therapy (none, chemotherapy, chemoradiotherapy)
5. Histology (squamous or adenocarcinoma).

All patients considered for the trial will have a proforma filled for pre, intra and postoperative details (Annexure 4). Preoperative patient preparation would be routine and identical in both groups and will include chest physiotherapy, deep breathing exercises and incentive spirometry. Bronchodilators and antibiotics will be used selectively only if indicated.

Trial schema Patients with esophageal cancer

Staging investigations (CT scan, EUS, FOB) indicating operable disease with surgical plan of total transthoracic esophagectomy

Investigations for fitness for surgery indicating good risk for surgery STRATIFY

1. Preoperative T stage (T1&2, T3 and T4)
2. Preoperative N stage (N0, N1)
3. Level of disease (upper, middle and lower third)
4. Neoadjuvant therapy (none, chemotherapy, chemoradiotherapy)
5. Histology (squamous or adenocarcinoma)

RANDOMIZE

Three field esophagectomy Two field esophagectomy

All surgeries will be performed under general anesthesia with epidural analgesia. The surgery will be either performed by or under the direct supervision of consultant thoracic surgeons with experience in esophageal surgery. Thoracic esophageal mobilization and mediastinal lymphadenectomy will be done by open thoracotomy or video assisted thoracoscopic surgery. Lymphadenectomy will be as defined in the consensus conference of the fifth IGSC at Munich.

Field 1. The abdominal field will include all lymphatic and connective tissues between the hiatus cranially, the upper border of the pancreas caudally, the splenic hilum to the left and the hepatoduodenal ligament and right gastric artery to the right.

Field II. This refers to the intrathoracic compartment and is defined as

1. Standard lymphadenectomy: This includes para esophageal lymph nodes, subcarinal lymph nodes and right and left para bronchial lymph nodes.
2. Extended lymphadenectomy: This includes the standard lymphadenectomy plus the right apical nodes, right recurrent nerve nodes and the right paratracheal nodes.
3. Total lymphadenectomy: This includes the extended lymphadenectomy plus the left apical nodes plus the left recurrent nerve and paratracheal nodes.

Field III. This refers to the cervical compartment and includes clearance in the omohyoid triangle with sparing of the sternocleidomastoid muscle and the internal jugular vein. The cranial landmark is the cricoid cartilage and the caudal landmark the upper margin of the clavicle.

Three-field lymphadenectomy: The type of resection will include lymph node clearance of Fields I and III and a total type Field II lymphadenectomy.

Two field lymphadenectomy: The type of resection will include lymph node clearance of Field I and any of the types of lymphadenectomy in Field II. Standard mediastinal lymphadenectomy will be done in all patients; no special effort will be made to dissect the supracarinal compartment unless grossly enlarged lymph nodes are seen.

Three field lymphadenectomy Two field lymphadenectomy

Operative time, blood loss, blood product replacement and all intraoperative details will be recorded in the proforma. Patients will be shifted postoperatively to the intensive care unit (ICU) for observation and subsequently to the recovery or high dependency ward once stabilized. Postoperative details including period of postoperative ventilation, hemorrhage, pulmonary and cardiac complications, arrhythmias, thoracic duct leak, anastomotic leak, wound infection and recurrent laryngeal nerve paresis or palsy will be recorded. Postoperative complications will be recorded as per Annexure 5. Postoperative mortality will be defined as 30-day mortality plus death before discharge after surgery.

Patients will be started on oral feeds between the 8th and 10th day in the absence of an anastomotic leak. The total duration of ICU stay and hospital stay will also be recorded.

Follow up Patients will be followed up four to six monthly for the first three years and annually thereafter. A detailed history and clinical examination will be done on every follow up with the quality of speech, swallowing recorded. Patients who had a fixed cord postoperatively will undergo laryngoscopy to assess recovery of function. Symptomatic patients will be investigated by upper gastrointestinal endoscopy, CT scan, ultrasound and haematological and biochemical investigations. Asymptomatic patients will not be routinely investigated.

Sample size The sample size considering an improvement of survival from 25% to 35% will be 588 patients (289 in each arm). The trial will aim at enrolling 700 patients in order to adjust for loss to follow up and protocol violations. Interim analyses will be done when ¼ th (103 events) and ½ (206 events) of the estimated events occur. We expect to complete accrual of patients in seven years.

Data management All collected data will be entered into a statistical software package for subsequent analysis (SPSS for Windows, Version 11.5)

Main research variables Primary end point Overall survival in the two arms Secondary endpoints

1. Disease free survival
2. Locoregional recurrence
3. Postoperative morbidity and mortality
4. Quality of life - short and long term

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy or cytology proven (squamous or adenocarcinoma) esophageal cancer
* Patients with staging investigations showing operability
* Surgical plan of total transthoracic esophagectomy

Exclusion Criteria:

* Patients with low performance status (ECOG score>1)
* Past history of malignancy
* Staging investigations indicating advanced disease
* Patients medically unfit for surgical resection
* Patients with pulmonary reserve inadequate to undergo thoracotomy and extensive mediastinal lymphadenectomy
* Patients considered for salvage surgery after definitive (radical)chemoradiotherapy
* Patients with supracarinal lymph node enlargement on CT scan and/or EUS
* Patients intraoperatively detected to have grossly enlarged supracarinal lymph nodes
* Patients with Siewert's type III CO junction growths
* Patients above the age of 70 years
* Patients unreliable for follow up

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700
Dates: Start 2005-01; Study Completion 2015-12

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Disease-free survival
Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh C Mistry, MS, Principal Investigator — Tata Memorial Hospital; C S Pramesh, MS, FRCS, Principal Investigator — Tata Memorial Hospital
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India